CLINICAL TRIAL: NCT07003802
Title: The Contributions of Neural Control and Mechanosensation to Rehabilitation Induced Spine Muscle Recovery
Brief Title: Neural Control and Mechanosensation in Spine Muscle
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Bahar Shahidi, Associate Professor, University of California, San Diego
Other Study IDs: HD088437-06
Record Dates: First submitted 2025-05-20; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain and Core Muscle; Disc Herniation
Keywords: low back pain; exercise; physical therapy; surgery
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — paraspinal muscle biopsies from individuals undergoing surgery for lumbar spine pathology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Physical Therapy cohort: Individuals who have been prescribed and are initiating an exercise based physical therapy program for their low back pain
  Interventions: Behavioral: Resistance exercise
- Surgical Cohort: Individuals who are undergoing surgical management for chronic disc disease
  Interventions: Behavioral: Resistance exercise
- Healthy Cohort: Individuals with no history of low back pain or pathology
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Resistance exercise — An acute bout of a 3 minute resistance exercise will be performed using a lumbar extension exercise machine

SUMMARY:
Low back pain (LBP) is a condition that affects a majority of the US population and is responsible for a significant proportion of health care costs and utilization. Lumbar spine muscle is compromised in LBP, and do, and do not, respond to exercise based physical therapy program depending on measurements representing activation capacity of lumbar muscle. Here, we will characterize the neurological and muscle specific features that may contribute to limited activation in an attempt to identify sources of resistance to recovery in patients with chronic disc injury and identify precision rehabilitation approaches for this complex population of individuals.

DETAILED DESCRIPTION:
Low back pain (LBP) is a complex condition that affects 65-85% of the population, and is the leading musculoskeletal condition contributing to disability in the United States. Disc injury is the most common injury and 75% of individuals undergoing surgical and rehabilitative interventions for this condition experience suboptimal or poor outcomes. These patients demonstrate disability and deficits in functional capacity, and paraspinal muscles in these individuals have been shown to be altered in volume, composition, and mechanical properties. These maladaptive changes influence the ability for the muscle to respond appropriately to rehabilitation efforts in a subgroup of individuals with chronic back pain who do not demonstrate the expected acute activation responses to exercise. While the structural and adaptive capacities of healthy muscle are well understood, pathological muscle recovery and activation deficits are less clear and may be influenced by neurogenic and/or muscle specific impairments. To address this gap in knowledge, the purpose of this trial is to compare central and peripheral origins of impaired activation in individuals with chronic disc injury who do, and do not respond to exercise. Experiment 1 will use a novel functional MRI technique and electromyographic measurements to compare responder and non-responder groups in patients with chronic lumbar disc injury undergoing standard physical therapy. Experiment 2 will compare corticomotor excitability and intracortical inhibition and facilitation between individuals who are undergoing physical therapy or surgery who do and do not respond to exercise. Experiment 3 will compare ex vivo passive and active mechanical responses, and transcriptomics from intraoperative multifidus biopsies of patients undergoing spinal surgery for chronic lumbar disc injury to evaluate muscle mechanotransduction. These experiments will elucidate the neurogenic and muscle-specific contributions to muscle adaptation in the presence of chronic lumbar spine pathology and pain.

ELIGIBILITY:
Inclusion Criteria:

* Surgical group:
* Individuals diagnosed with chronic disc injury (symptoms > 3 months),
* Individuals planning to undergo a spinal surgery to address the diagnosis of chronic disc injury

Physical Therapy Group-

* Individuals diagnosed with chronic disc injury (symptoms >3 months),
* Individuals initiating an exercise-based physical therapy program to address the diagnosis of chronic disc injury

Healthy Control group -

* Individuals with no history of chronic back pain (interfering pain lasting >3 months) within the past 3 years,
* no significant spinal pathology beyond normal age-related degenerative changes

Exclusion Criteria:

* Surgery/Physical therapy groups-History of lumbar spine surgery
* Diabetes
* Neuromuscular diseases
* Epilepsy or other seizure disorder -Healthy control group -
* History of lumbar spine surgery
* History of interfering pain lasting >3 months
* Diabetes
* Neuromuscular diseases
* Epilepsy or other seizure disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Disc Injury or Healthy Control
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2031-04-01 (Estimated); Study Completion 2033-04-01 (Estimated)

PRIMARY OUTCOMES:
RMS amplitude of paraspinal muscle EMG | Baseline
  Average RMS EMG amplitude of the lumbar multifidus over the duration of the acute exercise bout.
IVIM responsiveness | Baseline
  Response classification from IVIM MRI imaging as an increase in IVIM Diffusion (D) of at least 0.055 x 10-3 mm2/s and a pseudodiffusion (D*) increase of at least 6.94 x 10-3 mm2/s in response to the acute exercise stimulus
Cortical excitability | Baseline
  Transcranial Magnetic Stimulation based motor threshold of activation of the lumbar multifidus muscle
pAMPK | Time of surgery/biopsy
  Mechanically-induced phosphorylation of p38 MAPK-Thr180/Tyr182 (p-p38T180/Y182) from intraoperative multifidus biopsies or biopsy needle

SECONDARY OUTCOMES:
MEP amplitude | Baseline
  Motor evoked potential of multifidus in response to Transcranial Magnetic Stimulation of the motor cortex
Cortical Silent Period | Baseline
  Period of motor silence in the multifidus after Transcrianial Magnetic Simulation MEP over the motor cortex
Short Interval Intracortical Inhibition (SICI) | Baseline
  Measurement of signal loss in the multifidus after a paired pulse stimulation of the motor cortex using transcranial magnetic stimulation
Short Interval Intracortical Facilitation (SICF) | Baseline
  Measurement of time of multifidus muscle activation after a paired pulse transcranial magnetic stimulation of the motor cortex
p-mTORS2448/total mTOR | Time of surgery/biopsy
  Structural Proteins and phosphorylation of p-mTORS2448/total mTOR measured from intraoperative multifidus biopsies or biopsy needle

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
10 channel EMG data, 2 channel TMS data, MRI images, and biopsy-based signaling and sequencing data
Supporting Information: Study Protocol, Analytic Code

DOCUMENTS (1):
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT07003802/ICF_000.pdf